CLINICAL TRIAL: NCT03341221
Title: Diagnosis of Ascites in Infants and Children
Acronym: Ascites
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa abo bakr Ahmed, Doctor, Assiut University
Other Study IDs: Assuit university 246810
Record Dates: First submitted 2017-10-28; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group: Diagnosis of ascites in infants and children by history, examination and investigations

SUMMARY:
Ascites is the pathologic accumulation of fluid within the peritoneal cavity. Causes of ascites in infants and children :hepatobiliary disorders,serositis, neoplasm, cardiac, genitourinary disorder, metabolic disease and others.

Diagnosis of ascites :history of abdominal distention, increasing weight, respiratory embarrassement, symptoms and signs of (hepatic ,cardiac,renal disease, tuberculosis and malignancy).

lnvestigation:complete blood count, complete urine examination, liver function tests, plasma proteins, renal function tests, clotting screen, tuberculin test, chest and abdominal plain films,abdominal ultrasound, upper gastrointestinal endoscopy, abdominal paracentesis for ascitic fluid analysis .

DETAILED DESCRIPTION:
Definition : Ascites is the pathologic fluid accumulation within the peritoneal cavity .

causes of ascites in infants and children :

* Hepatobiliary disorders (cirrhosis, congenital hepatic fibrosis, acute hepatitis B,C ,Budd -chiari syndrome, Bile duct perforation)
* Serositis (crohn's disease, eosinophilic enteropathy , Henoch- Shonlein purpura )
* Neoplasm (lymphoma, wilm's tumor ,Glioma, Germ cell tumor, Ovarian tumor,mesothelioma, Neroblastoma )
* Cardiac (Heart failure )
* Metabolic disease
* Gastrointestinal disorder (Nephrotic syndrome, peritoneal dialysis ). Diagnosis of ascites :History of abdominal distention, increasing weight, respiratory embarrassement, jaundice, bleeding (haematemsis, melena, and epistaxis ),Pruritus ,Growth failure ,abdominal pain, fever,Cyanosis, ,dyspnea during suckling, Orthopnea, Buffy eyes, lower limb swelling, Haematrruria .

By examination : Tachycardia ,Tachypnea ,Hypertension ,cyanosis, jaundice, clubbing of fingers ,limb edema ,Hepatomegaly, splenomegaly, dilated abdominal wall veins.

Investigations :

Laboratory tests :complete blood count , complete urine examination, liver function tests, plasma proteins, renal function tests, clotting screen, tuberculin test.

Imaging studies :chest and abdominal plain films, abdominal ultrasound, upper gastrointestinal endoscopy CT, MR I, Abdominal paracentesis for ascitic fluid analysis :cell count / cytology ,Gram 'stain and culture, Total proteins (albumin /globulin ratio ), Glucose, Amylase, lactase dehydrogenase, Triglycerides,Bilirubin.

Serum ascites albumin gradient (SAAG )is the best single test for classification of ascites into portal hypertensive (SAAG >1.1g/dl) and non-portal hypertensive (SAAG <1.1g/dl) causes.

ELIGIBILITY:
Inclusion Criteria:

* age from 1month to 18 year
* infants and children with ascites (hepatic, cardiac, renal, malignant or tuberculous )
* infants and children with peritonitis

Exclusion Criteria:

* age <1month
* surgical conditions as ruptured viscous or located abscess

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants and children with ascites aged from 1month to 18 year
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of ascites in infants and children with hepatic, cardiac, renal disease, tuberculosis and malignancy | 1 year
  Diagnosis of ascites in infants and children fromega age of 1month to 18 year